CLINICAL TRIAL: NCT04355702
Title: Manifestations Related to Covid-19 in Patients With Systemic Lupus Erythematosus
Brief Title: Covid-19 in Lupus Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0219
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Systemic Lupus Erythematosus; Covid-19
Keywords: Systemic lupus erythematosus; Hydroxychloroquine
MeSH Terms: conditions — Lupus Erythematosus, Systemic; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lupus patients treated by hydroxychloroquine: Lupus patients treated by hydroxychloroquine
- Lupus patients not treated by hydroxychloroquine: Lupus patients not treated by hydroxychloroquine

SUMMARY:
The Covid-19 pandemic is a major public health issue. Potential treatments are essential to control the infection. Hydroxychlorquine is currently tested in several clinical trials to evaluate its efficiency.The objective of this study was to evaluate the symptoms related to COVID-19 occuring in patients with systemic lupus erythematosus (SLE)

DETAILED DESCRIPTION:
Introduction:The Covid-19 pandemic has had a major impact on many countries on the sanitary and economic level. Finding an efficient cure is paramount in order to reduce its severity and mortality. Several medications are currently under investigation. Among them, hydroxychloroquine can prevent viral replication at several sites and has been shown efficient in vitro. Several clinical trials are in progress to evaluate its efficiency in vivo. However, no study so far has evaluated the covid-19 infection in patients with SLE.

Objectives and methods: The primary objective was to describe the prevalence and the severity of Covid-19 infection in patients wih systemic lupus erythematosus. The secondary objective was to compare these parameters in patients treated by hydroxychloroquine and those not treated by hydroxychloroquine. This observational study of a historical-prospective cohort focuses on all adult lupus patients seen during the last year in the departments of rheumatology and nephrology in CHU Montpellier. It will collect information concerning the patient's condition, treatments and main comorbidities (cardio-vascular, respiratory, hepatic and immune depression), as well as symptoms suggesting covid-19 infection, its confirmation and its course and severity.

ELIGIBILITY:
Inclusion criteria:

- adult patient with systemic lupus erythematosus seen during the last year in the departments of rheumatology or nephrology

Exclusion criteria:

- patient not speaking french nor english

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients with systemic lupus erythematosus followed by the departments of rheumatology and nephrology, seen during the last year
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
prevalence and severity of Covid-19 infection in patients with SLE | 1 day
  prevalence and severity of Covid-19 infection in patients with SLE

SECONDARY OUTCOMES:
prevalence and severity of Covid-19 infection in patients treated by hydroxychloroquine | 1 day
  prevalence and severity of Covid-19 infection in patients treated by hydroxychloroquine

CONTACTS AND LOCATIONS:
Overall Officials: Christian JORGENSEN, Resident, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC